CLINICAL TRIAL: NCT00553397
Title: Live Lung Donor Retrospective Study (RELIVE-02)
Brief Title: Live Lung Donor Retrospective Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: DAIT RELIVE-02; RELIVE
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Lung Transplantation
Keywords: Living donor lung transplant; End stage lung disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Live Lung Donors: Participants had a living donor lobectomy at one of the two participating study centers, the University of Southern California and the Washington University Medical Center between 1993 and 2006.

SUMMARY:
The use of live donors for solid organ transplantation has increased the number of available organs for those waiting for a transplant. Donation of an organ may have significant effects on a donor's health. This study will determine the baseline characteristics, early postoperative morbidity, and long-term survival for participants who underwent donor lobectomy between 1993 and 2006.

DETAILED DESCRIPTION:
As the number of patients requiring organ transplants continues to increase, the number of organs available from deceased donors cannot meet demands. Beginning in the early 1990s, organs from living donors became a widely-available option, increasing the number of available organs for transplant. However, because organ donation has the potential to adversely affect a living donor's health, long-term studies to determine the effect of donation on these donors are needed. The purpose of this study is to determine the mortality, the early postoperative morbidity, and the occurrence of end stage lung disease for participants who underwent donor lobectomy between 1993 and 2006. Participants in this study will have had donor lobectomy at the University of Southern California in Los Angeles or the Washington University Medical Center and Barnes-Jewish Hospital in St. Louis.

There will be no study visits for retrospective cohort study. Investigators will collect data from existing medical records and databases.

ELIGIBILITY:
Inclusion Criteria:

* Had living donor lobectomy at one of the two participating study centers, the University of Southern California and the Washington University Medical Center between 1993 and 2006 (inclusive)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults who have donated a lung at either the University of Southern California or Washington University between 1993 and 2006
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Overall Mortality | Year 5

SECONDARY OUTCOMES:
Perioperative morbid events /complications | Year 5
Cause of death | Year 5
Incidence of Donors Requiring Lung Transplantation | Year 5
  Incidence of any of the donors who encountered complications related to their donation, which eventually resulted in them receiving lung transplantations.

CONTACTS AND LOCATIONS:
Overall Officials: Akinlolu Ojo, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Washington University Medical Center, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Barr ML, Belghiti J, Villamil FG, Pomfret EA, Sutherland DS, Gruessner RW, Langnas AN, Delmonico FL. A report of the Vancouver Forum on the care of the live organ donor: lung, liver, pancreas, and intestine data and medical guidelines. Transplantation. 2006 May 27;81(10):1373-85. doi: 10.1097/01.tp.0000216825.56841.cd. No abstract available. PMID 16732172
- [Background] Barr ML, Schenkel FA, Cohen RG, Barbers RG, Fuller CB, Hagen JA, Wells WJ, Starnes VA. Recipient and donor outcomes in living related and unrelated lobar transplantation. Transplant Proc. 1998 Aug;30(5):2261-3. doi: 10.1016/s0041-1345(98)00612-5. No abstract available. PMID 9723463
- [Background] Battafarano RJ, Anderson RC, Meyers BF, Guthrie TJ, Schuller D, Cooper JD, Patterson GA. Perioperative complications after living donor lobectomy. J Thorac Cardiovasc Surg. 2000 Nov;120(5):909-15. doi: 10.1067/mtc.2000.110685. PMID 11044317
- [Background] Bowdish ME, Barr ML. Living lobar lung transplantation. Respir Care Clin N Am. 2004 Dec;10(4):563-79. doi: 10.1016/j.rcc.2004.06.004. PMID 15585183
- [Background] Bowdish ME, Barr ML, Schenkel FA, Woo MS, Bremner RM, Horn MV, Baker CJ, Barbers RG, Wells WJ, Starnes VA. A decade of living lobar lung transplantation: perioperative complications after 253 donor lobectomies. Am J Transplant. 2004 Aug;4(8):1283-8. doi: 10.1111/j.1600-6143.2004.00514.x. PMID 15268729
- [Background] Goldsmith MF. Mother to child: first living donor lung transplant. JAMA. 1990 Dec 5;264(21):2724. No abstract available. PMID 2232048
- [Background] Mallory GB Jr, Cohen AH. Donor considerations in living-related donor lung transplantation. Clin Chest Med. 1997 Jun;18(2):239-44. doi: 10.1016/s0272-5231(05)70375-0. PMID 9187818
- [Background] Shaw LR, Miller JD, Slutsky AS, Maurer JR, Puskas JD, Patterson GA, Singer PA. Ethics of lung transplantation with live donors. Lancet. 1991 Sep 14;338(8768):678-81. doi: 10.1016/0140-6736(91)91244-o. No abstract available. PMID 1679484
- [Background] Starnes VA, Barr ML, Schenkel FA, Horn MV, Cohen RG, Hagen JA, Wells WJ. Experience with living-donor lobar transplantation for indications other than cystic fibrosis. J Thorac Cardiovasc Surg. 1997 Dec;114(6):917-21; discussion 921-2. doi: 10.1016/S0022-5223(97)70005-9. PMID 9434686
- [Result] Yusen RD, Hong BA, Messersmith EE, Gillespie BW, Lopez BM, Brown KL, Odim J, Merion RM, Barr ML; RELIVE Study Group. Morbidity and mortality of live lung donation: results from the RELIVE study. Am J Transplant. 2014 Aug;14(8):1846-52. doi: 10.1111/ajt.12771. PMID 25039865
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: National Heart, Lung, and Blood Institute (NHLBI) website — https://www.nhlbi.nih.gov/
- Available data/document: Individual Participant Data Set: SDY293 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY293 — ImmPort study identifier is SDY293
- Available data/document: Study Protocol: SDY293 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY293 — ImmPort study identifier is SDY293. The study protocol is available in the Design tab section.
- Available data/document: Study summary, -design, -demographics, -files: SDY293 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY293 — ImmPort study identifier is SDY293